CLINICAL TRIAL: NCT01610622
Title: Estimation of Cardiac Output in Neonatal ICU Using an Ultrasound Dilution Technique
Acronym: CH
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-COSTATUS-4A-H; R44HL061994 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Neonatal Intensive Care
Keywords: Cardiac Output; Blood volumes; Neonates

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: COstatus cardiac output measurement with isotonic saline — Isotonic saline, which is the indicator, is injected to obtain COstatus cardiac output measurements.
  No other interventions are made for the purpose of the study.

SUMMARY:
Presently there is no apparatus, clinically available, for routine determination of cardiac output (CO) in children. The goal of this research is to develop new technology that will help determine CO in neonates.

ELIGIBILITY:
Inclusion Criteria:

* All neonatal patients cared for in our ICU with umbilical venous and arterial catheters simultaneously in place for their care, will be eligible.

Exclusion Criteria:

* Patients would be excluded if the family/guardian denied permission or if the attending physician felt the patient was not stable.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Marr, MD, Principal Investigator — Crouse Hospital
Locations (1):
- Crouse Hospital, Syracuse, New York, United States